CLINICAL TRIAL: NCT06797219
Title: Light Therapy Device for Neonatal Intraventricular Hemorrhage Grade 3 and 4
Acronym: EFIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Onajovwe Fofah, MD, Department of Pediatrics Chair, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2023001886
Record Dates: First submitted 2024-08-06; First posted 2025-01-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Intraventricular Hemorrhage of Prematurity; Hydrocephalus
Keywords: low level laser therapy; neonate; developmental milestones; intraventricular hemorrhage
MeSH Terms: conditions — Hydrocephalus | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: A device to promote resorption and recovery from intraventricular hemorrhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Non-blinded, open label experimental arm (Experimental): The experimental arm will be administered treated with the study device. It will be 10 mW/cm^2 of 650nm laser through use of a novel laser device given for 5 minutes twice daily for 12 days.
  Interventions: Device: Low Level Laser Therapy for Intraventricular Hemorrhage of Prematurity

INTERVENTIONS:
Device: Low Level Laser Therapy for Intraventricular Hemorrhage of Prematurity — The experimental arm will be administered treated with the study device. It will be 10 mW/cm^2 of 650nm laser through use of a novel laser device given for 5 minutes twice daily for 12 days.

SUMMARY:
The primary purpose of this study is to serve as a pilot study of the EFIL device treatment feasibility of IVH grades 3,4 to guide development of a larger trial. Primary outcomes will assess the following: safety of intervention, recruitment and consent process, acceptability of intervention by parents, retention rates, selection of most appropriate outcome measures, provide sample size estimates for a larger trial, increase the researchers' experience with the study intervention. A complete list of objectives and aims are listed under "Objectives". This study hopes to treat 12-24 neonates using 650nm light of irradiance 10mW/cm2 for 5 minutes twice a day each day for 12 days. We will also call the parents at 6 months and 12 months to track developmental milestones.

ELIGIBILITY:
Inclusion Criteria:

* neonates with intraventricular hemorrhage grade 3 or 4 less than 1 month old.

Exclusion Criteria:

* neonates without IVH grade 3/4 or older than 1 month.

Ages: 0 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage Resorption Rate | Hemorrhage resorption rate tracking starts from date of identified intraventricular hemorrhage on head ultrasound (usually within 1 week of life) and head ultrasounds weekly up to 4 months old
  Measure rate at which neonate intraventricular hemorrhage is resorbed via serial head ultrasounds
Anterior Horn Width | Ventricle volume tracking starts from date of identified intraventricular hemorrhage on head ultrasound (within 1 week of life) performed through weekly head ultrasounds up to 4 months old
  Measure rate at which neonate intracranial pressure changes using anterior horn width (mm) derived from serial head ultrasounds.
Neurosurgical Interventions | Number of neurosurgical interventions starts at birth and continues up to 4 months old
  number of patients requiring neurosurgical intervention
Neurodevelopmental Outcomes at 6 months and 12 months of age | Two time points at 6 months of age and 12 months of age
  A phone survey will be conducted inquiring which developmental milestones have been met at 6 months (i.e., sitting independently, reaching to grab toys, knows familiar people, takes turns making sounds with care giver) and 12 months (plays interactive games, says mama/dada, looks for hidden objects, cruises, pincer grasp)
Ventricular Index | Ventricle volume tracking starts from date of identified intraventricular hemorrhage on head ultrasound (within 1 week of life); and subsequent weekly head ultrasounds performed up to 4 months old
  Measure rate at which neonate intracranial pressure changes using ventricular index (mm) derived from serial head ultrasounds.
Head Circumference | Head Circumference tracking starts from birth and is performed daily up to 4 months old
  Measure rate at which neonate intracranial pressure changes via head circumference (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Onajovwe Fofah, Medical, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Rutgers - New Jersey Medical School / University Hospital, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li D, Liu S, Yu T, Liu Z, Sun S, Bragin D, Shirokov A, Navolokin N, Bragina O, Hu Z, Kurths J, Fedosov I, Blokhina I, Dubrovski A, Khorovodov A, Terskov A, Tzoy M, Semyachkina-Glushkovskaya O, Zhu D. Photostimulation of brain lymphatics in male newborn and adult rodents for therapy of intraventricular hemorrhage. Nat Commun. 2023 Sep 29;14(1):6104. doi: 10.1038/s41467-023-41710-y. PMID 37775549
- [Background] Zivin JA, Albers GW, Bornstein N, Chippendale T, Dahlof B, Devlin T, Fisher M, Hacke W, Holt W, Ilic S, Kasner S, Lew R, Nash M, Perez J, Rymer M, Schellinger P, Schneider D, Schwab S, Veltkamp R, Walker M, Streeter J; NeuroThera Effectiveness and Safety Trial-2 Investigators. Effectiveness and safety of transcranial laser therapy for acute ischemic stroke. Stroke. 2009 Apr;40(4):1359-64. doi: 10.1161/STROKEAHA.109.547547. Epub 2009 Feb 20. PMID 19233936
- [Background] Naeser MA, Saltmarche A, Krengel MH, Hamblin MR, Knight JA. Improved cognitive function after transcranial, light-emitting diode treatments in chronic, traumatic brain injury: two case reports. Photomed Laser Surg. 2011 May;29(5):351-8. doi: 10.1089/pho.2010.2814. Epub 2010 Dec 23. PMID 21182447
- [Background] Huisa BN, Stemer AB, Walker MG, Rapp K, Meyer BC, Zivin JA; NEST-1 and -2 investigators. Transcranial laser therapy for acute ischemic stroke: a pooled analysis of NEST-1 and NEST-2. Int J Stroke. 2013 Jul;8(5):315-20. doi: 10.1111/j.1747-4949.2011.00754.x. Epub 2012 Feb 2. PMID 22299818
- [Background] Lampl Y, Zivin JA, Fisher M, Lew R, Welin L, Dahlof B, Borenstein P, Andersson B, Perez J, Caparo C, Ilic S, Oron U. Infrared laser therapy for ischemic stroke: a new treatment strategy: results of the NeuroThera Effectiveness and Safety Trial-1 (NEST-1). Stroke. 2007 Jun;38(6):1843-9. doi: 10.1161/STROKEAHA.106.478230. Epub 2007 Apr 26. PMID 17463313
- [Background] Kent AL, Broom M, Parr V, Essex RW, Abdel-Latif ME, Dahlstrom JE, Valter K, Provis J, Natoli R. A safety and feasibility study of the use of 670 nm red light in premature neonates. J Perinatol. 2015 Jul;35(7):493-6. doi: 10.1038/jp.2015.5. Epub 2015 Feb 19. PMID 25695843